CLINICAL TRIAL: NCT04606862
Title: A Non-Randomized Clinical Trial to Investigate the Efficacy of the Morley Medical Sepsis (MMS) Software Device in the Prediction and Early Detection of Sepsis
Brief Title: A Clinical Trial to Evaluate the Efficacy of the Morley Medical Sepsis (MMS) Software Device in Predicting Sepsis in Adult Patients Using Artificial Intelligence (AI) Machine Learning Algorithms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Morley Medical (Industry)
Collaborators: Morley Research Consortium (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MMSEP1901
Record Dates: First submitted 2020-10-21; First posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Intervention Model Description: This is a pivotal medical device clinical trial comparing the clinical outcomes in hospitalized patients monitored with the MMS Software Device for the prediction and early detection of sepsis versus patients monitored with current standard sepsis scoring systems at participating clinical trial sites. This will be conducted through a non-randomized multi-center, non-blinded, clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Investigational Arm (Experimental): The patients enrolled into the investigational arm at each participating hospital will be monitored with the Morley Medical Sepsis (MMS) Software Device for the prediction and early identification of sepsis.
  Interventions: Device: Morley Medical Sepsis Software Device
- Control Arm (No Intervention): The patients enrolled into the control group of each participating hospital will not be monitored with the Morley Medical Sepsis (MMS) Software Device for the prediction and early identification of sepsis. These patients will be monitored according to each institution's standard sepsis screening practices.

INTERVENTIONS:
Device: Morley Medical Sepsis Software Device — The Morley Medical Sepsis (MMS) Software Device is a predictive analytics, stand-alone, cloud-based software system with no hardware components. The software acquires patient data from the electronic medical record, processes the data using unique artificial intelligence (AI) powered algorithms, and generates clinical decision support outputs that aid in the proactive delivery of customized and efficient care for patients. The software output is made available to the end users (trained medical professionals) via an intuitive user interface displayed on desktop computers or mobile communication devices such as laptops, smartphones or tablets.
  Arms: Investigational Arm

SUMMARY:
This is a pivotal medical device clinical trial evaluating the clinical outcomes in hospitalized patients monitored with the Morley Medical Sepsis Software Device. The device uses unique AI machine learning algorithms to analyze patient data in real time and generate clinical decision support sepsis risk predictions for clinicians.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient 18 years of age or older
* Patient is admitted or had been admitted to a participating healthcare facility

Exclusion Criteria:

* Sepsis diagnosis present on admission
* Involvement in a clinical trial of another investigational product with similar purpose

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2020-10-31 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
In-hospital sepsis prevalence | Up to 8 weeks
In-hospital sepsis related 30-day mortality | 30 days

SECONDARY OUTCOMES:
In-hospital all-cause 30-day mortality | 30 days
Hospital length of stay | Up to 8 weeks
Hospital re-admission | Up to 8 weeks
Time of initial IV fluids administration | Day 1 to Day 30, or until discharge
Time of initial vasopressors administration | Day 1 to Day 30, or until discharge
Time of initial antibiotics administration | Day 1 to Day 30, or until discharge
Time of initial blood microbiology culture | Day 1 to Day 30, or until discharge
Sepsis related adverse outcomes (septic shock) | Day 1 to Day 30, or until discharge
Sepsis prediction to onset time | Day 1 to Day 30, or until discharge
Sensitivity and specificity of sepsis prediction | Day 1 to Day 30, or until discharge